CLINICAL TRIAL: NCT01724879
Title: Open Label Phase II Study to Evaluate the Safety of Standard Induction and Consolidation Therapy in Combination With Dasatinib in Newly Diagnosed Adult Patients With Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (PH+ALL)
Brief Title: Study of Frontline Dasatinib Plus Chemotherapy in Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (PH+ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, MD, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL-PH-01; 2010-022854-18 (EudraCT Number)
Record Dates: First submitted 2012-02-03; First posted 2012-11-12 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Philadelphia Positive Acute Lymphoblastic Leukemia
Keywords: philadelphia chromosome; BCR-ABL; ALL; acute lymphoblastic leukemia; dasatinib; Sprycel
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia Chromosome | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib and chemotherapy (Experimental): Dasatinib, QD p.o. administration, day 1 to EOS
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Dasatinib p.o. + Chemotherapy (Dexamethasone, Cyclophosphamide, Vincristine, Methotroxate, 6-Mercapto-Purine, Cytarabine, Vindesine, VP16 (Etoposide))
  Other Names: Sprycel (R); BMS-354825

SUMMARY:
The current standard treatment approach for young patients with Positive Acute Lymphoblastic Leukemia (Ph+ALL) is the combination of a chemotherapy protocol employing four to five cytotoxic agents typically used for ALL together with imatinib. It is recommended to propose allogeneic Standard Induction and Consolidation Therapy (SCT) to all eligible patients with a suitable donor and to continue imatinib with or without additional therapy in patients not undergoing SCT.

This protocol is a study for newly diagnosed Philadelphia chromosome positive acute lymphoblastic leukemia in patients aged 18 to 55 years.

The objective of this strategy is to improve the overall results in the treatment of adult ALL with the addition of specific molecules to the common chemotherapeutic schedule.

DETAILED DESCRIPTION:
In the present study, the potent ABL tyrosine kinase inhibitor, Dasatinib will be added to standard induction and consolidation chemotherapy for the Philadelphia positive chromosome sub-group of ALL patients aged 18 to 55 years.

The Study hypothesis is, that Dasatinib in combination with standard chemotherapy according to GMALL protocol 07/2003 is feasible and induces cytologic and molecular remission rates comparable to chemotherapy in combination with imatinib without increased treatment-related mortality.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed new diagnosis of Philadelphia chromosome or BCR-ABL positive acute lymphoblastic leukemia
* Male or female patients aged 18-55 years
* Not previously treated except for prephase (corticosteroids, cyclophosphamide, single dose VCR will be permitted) therapy during establishment of the diagnosis
* Signed written inform consent, willingness and ability to comply with all study procedures
* Molecular detection of BCR-ABL transcripts
* Willingness of women of child-bearing potential (WOCBP) and male subjects whose sexual partners are WOCBP, to use an effective form of contraception (pearl index < 1%), such as complete sexual abstinence, combined oral contraceptive, hormone IUCD, vaginal hormone ring, transdermal contraceptive patch, contraceptive implant or depot contraceptive injection in combination with a second method of contraception like a condom or a cervical cap / diaphragm with spermicide or surgical sterilisation (vasectomy) in male patients or male partners during the study and at least 6 months thereafter. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or surgical sterilization or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months).
* Negative pregnancy test for women of child-bearing potential.

Exclusion Criteria:

* Patients with ECOG status > 2
* Patients with QTcF > 470 ms
* Cardiac insufficiency NYHA grade III/IV, LEVF < 50%, myocardial infarction within the past 6 months prior to study
* Active secondary malignancy requiring treatment
* Patients with active, uncontrolled bacterial, viral or fungal infection
* Known infection with HIV, Hepatitis B (except post vaccinal profile) or C
* Inadequate hepatic functions defined as ASAT or ALAT > 2,5 times the institutional upper limit of normal and total bilirubin > 2 fold the institutional upper limit unless considered to be due to organ involvement by the leukemia
* Concurrent severe diseases which exclude the administration of therapy
* Expected non-compliance or inability to understand informed consent
* Female patients who are pregnant or breast feeding
* Treatment with other investigational antileukemic agents after informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Treatment-related discontinuation of study treatment (Proportion of Patients) | Day 120

SECONDARY OUTCOMES:
Molecular complete remission rate (CR) | Day 120
Hematologic complete remission rate | Day 120
Grade III and IV txicity by Common Terminology Criteria for Adverse Events Version 3 | Day 120

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Gökbuget, Dr.med, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (22):
- Germany (22):
  - Robert Bosch Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Klinikum der Universität Regensburg, Regensburg, Bavaria
  - University Hospital of Frankfurt, Medical Dept. II, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinik Münster, Münster, North Rhine-Westphalia
  - Universitätsklinik Dresden, Dresden, Saxony
  - Uniklinik Aachen, Aachen
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinik Köln, Cologne
  - University Hospital Düsseldorf, Düsseldorf
  - Universitätsklinikum Göttingen, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Universität Leipzig, José-Carreras-Haus, Leipzig
  - Universitätskliniken Mainz, Mainz
  - Klinikum Mannheim, Mannheim
  - Universitätsklinikum Großhadern, München
  - Klinikum Nürnberg Nord, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Universität Rostock, Rostock
  - Medizinische Universitätsklinik Ulm, Ulm
  - Medizinische Poliklinik der Universität Würzburg, Würzburg